CLINICAL TRIAL: NCT05749237
Title: The Impact of Breath Exercises by Telemedicine in Patients Aged 8-18 Years With a Diagnosis of Asthma
Acronym: PHASTER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ayca Kiykim, Associate Professor, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Phaster
Record Dates: First submitted 2023-02-17; First posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Allergic Asthma
Keywords: allergy, asthma, respiratory exercises, children
MeSH Terms: conditions — Hypersensitivity; Asthma | interventions — Breathing Exercises

STUDY DESIGN:
Intervention Model Description: Randomized placebo controlled
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active group (Active Comparator): children older than 10 years with a diagnosis of allergic asthma respiratory and relaxation exercises
  Interventions: Other: respiratory exercises; Other: relaxation exercises
- Placebo group (Placebo Comparator): children older than 10 years with a diagnosis of allergic asthma only relaxation exercises
  Interventions: Other: relaxation exercises

INTERVENTIONS:
Other: respiratory exercises — respiratory exercises
  Arms: Active group
Other: relaxation exercises — relaxation exercises

SUMMARY:
The goal of this randomized, placebo controlled study is to evaluate the effect of respiratory exercises on asthma attack frequency, symptom and medication scores and quality of life of children with a diagnosis of asthma.

Participants will be asked to perform respiratory exercises described at once in hospital at home regularly. Control group will comprised children with asthma without respiratory exercises.

DETAILED DESCRIPTION:
At the beginning of the study anthropometric measurements, basal respiratory function assessment, drugs, demographic information, allergen sensitivity, asthma control levels and quality of life scales will be documented. Patients will be randomly divided into two groups; one group following respiratory exercises and relaxation exercises and the other following only relaxation exercises. Both groups will be called regularly to remind the exercises.

The spirometric tests and asthma control forms will be reevaluated at the 3rd and 6th month at hospital.

Peak flow meters will be given to patients to document PEF values during study.

ELIGIBILITY:
Inclusion Criteria:

clinical diagnosis of allergic asthma allergic asthma severity step 1 or step 2 -

Exclusion Criteria:

asthmatic children more severe than step 2 other comorbid disorders involving respiratory system or neuromusculatory disorders

-

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-03 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in asthma attack frequency | at third and sixth months
  asthma attack frequency by home PEF records and questionnaire, spirometric measurements and symptom and medication scoring charts

SECONDARY OUTCOMES:
Quality of life questionnaire | at third and sixth months
  increase quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Ayca Kiykim, Principal Investigator — Istanbul University - Cerrahpasa; Hilal Denizoglu, Study Chair — Atlas University; Hikmet Uçgun, Study Chair — Atlas University
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)